CLINICAL TRIAL: NCT01978483
Title: Effect of RANKL Inhibition on UV-induced Immunosuppression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Inno-6030
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Ultraviolet Rays; Immunosuppression; Hypersensitivity, Delayed; Immune Tolerance/Drug Effects
Keywords: Humans; Adult; skin; metabolism; radiation effects; Ultraviolet Rays; RANKL; RANK Ligand; denosumab; diphenylcyclopropenone; diphencyprone; immunology; immunosuppression; Antibodies, Monoclonal; Dermatitis, Allergic Contact; Hypersensitivity, Delayed
MeSH Terms: conditions — Hypersensitivity, Delayed; Dermatitis, Allergic Contact | interventions — Denosumab; RulB protein, Pseudomonas syringae; diphenylcyclopropenone; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- DPCP alone (Cohort 1) (Other): Diphenylcyclopropenone sensitization patches applied for 48hours. Diphenylcyclopropenone elicitation patches applied for 48hours.
  Interventions: Drug: Diphenylcyclopropenone
- UVB and denosumab group (Cohort 2) (Experimental): Denosumab 60mg subcutaneous injection once. Broadband UVB exposure once. Diphenylcyclopropenone sensitization patches applied for 48hours. Diphenylcyclopropenone elicitation patches applied for 48hours.
  Interventions: Drug: Denosumab; Radiation: UVB exposure; Drug: Diphenylcyclopropenone
- UVB and placebo group (Cohort 2) (Placebo Comparator): Normal saline 1mL subcutaneous injection once. Broadband UVB exposure once. Diphenylcyclopropenone sensitization patches applied for 48hours. Diphenylcyclopropenone elicitation patches applied for 48hours.
  Interventions: Radiation: UVB exposure; Drug: Diphenylcyclopropenone; Drug: Normal Saline

INTERVENTIONS:
Drug: Denosumab
  Other Names: Prolia
  Arms: UVB and denosumab group (Cohort 2)
Radiation: UVB exposure
  Other Names: Ultraviolet B rays; Ultraviolet B light
  Arms: UVB and denosumab group (Cohort 2); UVB and placebo group (Cohort 2)
Drug: Diphenylcyclopropenone
  Other Names: Diphencyprone; DPCP
Drug: Normal Saline
  Other Names: Saline 0.9%; NaCl solution 0.9%
  Arms: UVB and placebo group (Cohort 2)

SUMMARY:
Ultraviolet (UV) light is part of normal sunlight and has many effects on human skin and health. One of the harmful effects of long-term UV light exposure is that it can cause skin cancer. The mechanism by which UV light causes skin cancer is not entirely understood. One of the ways UV light causes cancer is by modifying DNA molecules in the cells of the skin. Another mechanism involved in cancer formation by UV light is immunosuppression. By this mechanism, UV light inactivates cells of the immune system of the skin. The immune cells are responsible for the detection and destruction of foreign substances and organisms such as bacterias and viruses but they also recognize and destroy cancer cells. UV light is known to prevent cells of the immune system to destroy cancer cells.

In laboratory experiments, a medication called denosumab has been shown to diminish the inhibition of ultraviolet-induced suppression of skin immunity. In other words, this medication could block the effect of UV on cells of the immune system and might allow patients taking this drug to be better protected from skin cancer.

The objective of this study is to test whether denosumab blocks the immunosuppressive effect of UVB light in healthy subjects. This study is divided into two stages. In the first stage, ten subjects (Cohort 1) will be sensitized to diphenylcyclopropenone (DPCP), a topical sensitizer commonly used for the treatment of alopecia areata and cutaneous warts. By reexposing the subjects to DPCP in incremental doses, dose-response levels of cutaneous hypersensitivity reactions in normal skin will be obtained. This will allow comparison of the normal levels of DPCP-induced cutaneous hypersensitivity (CHS) reaction in non UV-exposed skin (Cohort 1) to the CHS obtained from the two UVB-exposed experimental groups of Cohort 2.

In the second stage of the study, 20 subjects (Cohort 2) will be exposed to an immunosuppressive dose of ultraviolet B (UVB) 24 hours prior to DPCP sensitization. This is expected to result in the abolition of CHS upon rechallenge with DPCP. In order to assess whether denosumab can reverse UVB-induced immunosuppression, the subjects will have previously been randomized to receive a single 1mL injection of either 60 mg denosumab (group A; 10 subjects) or 1 mL saline (group B; 10 subjects) two weeks before UVB exposure. CHS reactions elicited by DPCP rechallenge will be compared between the denosumab and saline groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or postmenopausal women 18 years of age or older at time of consent.
* 2. Male subject or his female partner (this criterion does not apply to post-menopausal female) is willing to use effective contraceptive method for at least 30 days before Day 0 and at least 1 month after the last study drug administration. Effective contraceptive methods are:

  1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
  2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
  3. Intrauterine device (IUD);
  4. Sterilization such as tubal ligation, hysterectomy or vasectomy;
  5. Postmenopausal state for at least 1 year for female subject or female partner of male subject;
  6. Same-sex partner;
  7. Abstinence.
* 3. Capable of giving informed consent and the consent must be obtained prior to any study related procedures.
* 4. Fitzpatrick skin phototypes II or III.
* 5. Subject weighs 100kg or less.

Exclusion Criteria:

* 1. Conditions or medications causing immunosuppression, photosensitization or phototoxicity.
* 2. Past history of skin cancer or subject having precancerous skin lesions (eg. actinic keratosis).
* 3. Subject has atopic dermatitis (cohort 1)
* 4. Subject has received investigational drugs within the 28 days or 5 half-lives, whichever is longer, prior to Day 0 or plans to during the study period.
* 5. Subject has used any topical medication on arms or buttocks within 14 days of Day 0 or plans to during the study.
* 6. At the investigator's discretion subject has current or past history of alcohol or drug abuse that would interfere with the ability of the subject to comply with the study protocol.
* 7. Hypersensitivity/allergy to denosumab.
* 8. Hypersensitivity/allergy to lidocaine.
* 9. Hypersensitivity/allergy to latex.
* 10. Subject is taking anticoagulant medication except for low dose acetylsalicylic acid.
* 11. Past history of hypocalcemia or predisposing factors (eg, history of hypoparathyroidism, thyroid surgery, parathyroid surgery, malabsorption syndromes, excision of small intestine, severe renal impairment or receiving dialysis).
* 12. Known vitamin D deficiency.
* 13. Creatinine clearance less than 30mL/min (Cohort 2 only).
* 14. Corrected calcium concentration inferior to the normal range (Cohort 2 only).
* 15. Past history of osteonecrosis of the jaw (ONJ) or risk factors for ONJ (poor oral hygiene, periodontal and/or pre-existing dental disease, diagnosis of cancer with bone lesions, invasive dental procedures such as dental extractions or implants within 6 months of the screening visit.)
* 16. Past history of keloids or hypertrophic scarring.
* 17. Prior treatment with diphenylcyclopropenone.
* 18. Treatment with denosumab in the past 12 months.
* 19. Significant limitations in the range of motion of arms or shoulders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in dermal thickness: denosumab group vs placebo group of Cohort 2 | Three weeks after sensitization to DPCP.
  Mean dermal thickness, as measured by 20 MHz ultrasonography, after challenge with incremental doses of DPCP for subjects randomized to denosumab as compared to subjects randomized to placebo.

SECONDARY OUTCOMES:
Clinical score of contact hypersensitivity reactions: denosumab group vs placebo group of Cohort 2 | Three weeks after sensitization to DPCP.
  Mean clinical scores of contact hypersensitivity reaction sites elicited by incremental doses of DPCP challenges between the denosumab group and the placebo group.
Diameters of contact hypersensitivity reactions: denosumab group vs placebo group of Cohort 2 | Three weeks after sensitization to DPCP.
  Mean diameters (mm) of contact hypersensitivity reaction sites elicited by incremental doses of DPCP challenges between the denosumab group and the placebo group.
Change in dermal thickness: non UV-exposed (Cohort 1) vs UV-exposed (Cohort 2) | Three weeks after sensitization to DPCP.
  Mean dermal thickness, as measured by 20 MHz ultrasonography, after challenge with incremental doses of DPCP for subjects previously exposed to UVB as compared to subjects non-exposed to UVB.
Clinical score of contact hypersensitivity reactions: non UV-exposed (Cohort 1) vs UV-exposed (Cohort 2) | Three weeks after sensitization to DPCP.
  Mean clinical scores of contact hypersensitivity reaction sites elicited by incremental doses of DPCP between UV-exposed skin and non-UV exposed skin.
Diameters of contact hypersensitivity reactions: non UV-exposed (Cohort 1) vs UV-exposed (Cohort 2) | Three weeks after sensitization to DPCP.
  Mean diameters of contact hypersensitivity reaction sites elicited by incremental doses of DPCP between UV-exposed skin and non-UV exposed skin.
Gene expression levels: denosumab group vs placebo group of Cohort 2 | At baseline, two weeks after treatment injection, and 24 hours after UVB exposure.
  Differences in gene expression levels of RANK, RANKL and proteins that are regulated by the RANK-RANKL interaction in the denosumab versus placebo groups.
Histological pattern of expression of RANKL and other proteins of interest: denosumab group vs placebo group of Cohort 2 | At baseline, two weeks after treatment injection, and 24 hours after UVB exposure.
  Differences in the cutaneous histological pattern of expression of RANK, RANKL and proteins and cells that are involved in RANK-RANKL interaction in the denosumab versus placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada